CLINICAL TRIAL: NCT03441048
Title: A Phase I Study of Lintuzumab-Ac225 in Combination with CLAG-M Chemotherapy in Patients with Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Lintuzumab-Ac225 in Combination with Cladribine + Cytarabine + Filgastrim + Mitoxantrone (CLAG-M) for Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sameem M. Abedin, MD, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00031633
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Relapsed/refractory acute myeloid leukemia; CLAG-M; Lintuzumab
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Mitoxantrone; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Lintuzumab Ac225 (Dose 1 - 0.25 μCi/kg Ac-225 with 1.6 μg/kg lintuzumab) (Experimental): Dose escalation for lintuzumab-Ac225 will be conducted according to a 3+3 design. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF
- Lintuzumab Ac225 (Dose 2 - 0.50 μCi/kg Ac-225 with 3.2 μg/kg lintuzumab) (Experimental): Dose escalation for lintuzumab-Ac225 will be conducted according to a 3+3 design. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF
- Lintuzumab Ac225 (Dose 3 - 0.75 μCi/kg Ac-225 with 4.7μg/kg lintuzumab) (Experimental): Dose escalation for lintuzumab-Ac225 will be conducted according to a 3+3 design. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF
- Lintuzumab Ac225 (Dose 4 - 1.00 μCi/kg Ac-225 with 6.4 μg/kg lintuzumab) (Experimental): Dose escalation for lintuzumab-Ac225 will be conducted according to a 3+3 design. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF
- Lintuzumab Ac225 (Dose 5 - 1.25 μCi/kg Ac-225 with 8.0 μg/kg lintuzumab) (Experimental): Dose escalation for lintuzumab-Ac225 will be conducted according to a 3+3 design. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF
- Lintuzumab Ac225 Recommended Phase 2 Dose (RP2D) (Experimental): The maximum-tolerated dose for lintuzumab-Ac225 is defined as the highest level at which no more than one patient experiences a dose-limiting toxicity. The RP2D is defined as the dose level below the dose where two or more dose-limiting toxicities were observed. CLAG-M chemotherapy will be administered at a fixed dose and schedule (cladribine 5mg/m^2/day IV over two hours on days 2-6; cytarabine 2 gm/m^2/day IV over four hours on days 2-6, starting two hours after the cladribine infusion is complete; mitoxantrone 10mg/m^2/day IV on days 2-4 and G-CSF at a dose of 300 µg on days 1-6). Lintuzumab-Ac225 will be administered as a single dose on day 8 of therapy.
  Interventions: Biological: Lintuzumab-Ac-225; Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Drug: G-CSF

INTERVENTIONS:
Biological: Lintuzumab-Ac-225 — Lintuzumab-Ac225 is an immunoconjugate [antibody: anti-CD 33 antibody and radioactive isotope: Actinium (225Ac)] for the treatment of relapsed/refractory acute myeloid leukemia.
  Other Names: HuM195-Ac225; Actimab-A
Drug: Cladribine — Cladribine is a purine antimetabolite.
  Other Names: Leustatin; Mavenclad
Drug: Cytarabine — Cytarabine is an antineoplastic anti-metabolite.
  Other Names: Cytosar-U; Depocyt; cytosine arabinoside (ara-C)
Drug: Mitoxantrone — Mitoxantrone is an anthracenedione antineoplastic agent.
  Other Names: Mitozantrone; Novantrone
Drug: G-CSF — G-CSF is a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells.
  Other Names: colony-stimulating factor 3 (CSF 3)

SUMMARY:
This is a prospective, single-center phase I clinical study aimed at determining the maximum-tolerated dose, recommended phase 2 dose and safety of Lintuzumab-Ac225 in combination with CLAG-M chemotherapy in the management of relapsed/refractory acute myeloid leukemia. This study uses a 3+3 design with a five-patient cohort at the recommended phase 2 dose.

DETAILED DESCRIPTION:
Relapsed/refractory acute myeloid leukemia (RR-AML) in adults is an important therapeutic challenge. Nearly 60% of AML patients ultimately relapse or have refractory disease, and failure to achieve remission in this population is almost universally fatal. Therefore, a critical need exists for the development of novel therapies.

Currently, for RR-AML, many institutions utilize the chemotherapy regimen of CLAG-M (cladribine, cytarabine, G-CSF, mitoxantrone) based on a reported morphological complete remission (CR) rate of 58% in prospective clinical trials. Because of this, and its favorable performance when compared with outcomes reported for other regimens utilized in RR-AML, we believe enhancing the efficacy of CLAG-M is a rational approach to improve therapy in RR-AML.

A promising approach that could enhance the clearance of leukemic blasts when added to CLAG-M chemotherapy is a monoclonal antibody radioconjugate directed against markers expressed in leukemic cells. Radiation has known cytotoxic properties in chemo-resistant AML. The benefit of an antibody radioconjugate would be leukemic specific delivery of potent radiotherapy with potentially minimal systemic off-target side-effects. One such antibody radioconjugate is Lintuzumab-Ac225, a highly cytotoxic alpha radiation emitter that targets the cluster of differentiation 33 (CD33) cell surface antigen, which is expressed on leukemic cells.

In this novel study, we aim to add the radioconjugated antibody Lintuzumab-Ac225 to salvage CLAG-M chemotherapy in order to improve the treatment response for patients with RR-AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of informed consent.
2. Morphologically documented primary AML or secondary AML [from prior conditions such as Myelodysplastic Syndrome (MDS), myeloproliferative neoplasm (MPN)] or therapy related AML (t-AML), as defined by World Health Organization (WHO) criteria.
3. In first or subsequent relapse or refractory status after prior therapy, with or without prior hematopoietic stem cell transplant (HSCT). Patients with MDS and progression to AML on hypomethylating agents will also be included.
4. Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
5. Greater than 25% of blasts must be CD33 positive on flow cytometry using Phycoerythrin (PE) labeled anti-CD33 antibody.
6. Patients must meet the following clinical laboratory criteria:

   * Total bilirubin ≤ 2 x the upper limit of the normal range (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
   * Calculated creatinine clearance ≥ 50 mL/min
   * Resting left ventricular ejection fraction (LVEF) > 40%
7. Female patients must agree to avoid becoming pregnant, and male patients should avoid impregnating a female partner.

Exclusion Criteria:

1. Acute Promyelocytic Leukemia.
2. Active severe infection not well controlled by antibacterial or antiviral therapy.
3. Known infection with human immunodeficiency virus.
4. Patients with documented pulmonary disease, with a diffusing capacity of the lungs for carbon monoxide (DLCO) and/or forced expiratory volume in one second (FEV1) <65%, or history of dyspnea at rest, or requiring oxygen.
5. Pregnant or breast feeding women.
6. Prior chemotherapy or radiotherapy within 14 days of study entry unless fully recovered from adverse effects due to treatment, at investigator's discretion.
7. Active malignancy within 2 years of entry, except previously treated melanoma grade 2 or less, non-melanoma skin cancer, carcinoma in situ, or cervical intraepithelial neoplasia, and organ confined prostate cancer with no evidence of progressive disease based on prostate-specific antigen (PSA) levels and are not on active therapy. Active malignancy is malignancy receiving treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicities. | 28 Days
  Dose-escalation will be conducted according to a 3+3 design with a five-patient expansion cohort at the recommended phase 2 dose. The initial dose of Lintuzumab-Ac225 will be 0.25 micro-Curie (μCi)/kg (Dose level 1), and the highest dose administered will be 1.25 μCi/kg.
  * if 0/3 pts have no dose-limiting toxicity (DLT), new patients enter next dose level.
  * if 1/3 pts has DLT, 3 pts treated at same dose level.
  * if 0/3 pts at that dose level has DLT, new pts enter higher level.
  * if 1 or more of the additional 3 pts has a DLT, no further pts started at dose level, preceding dose is the MTD.
  * if 2/3 of initially dosed patients have a DLT on first dose, study terminated.
  * if 0/3 have DLT at highest dose, additional 3 enrolled.
Maximum-tolerated dose. | 28 Days
  Defined as the dosage with the highest level at which no more than one subject experiences a DLT.
The number of subjects who have at least one serious adverse event related to the study. | 60 days
  All subjects who receive study drug will be closely monitored for serious adverse events (SAEs). The NCI's CTCAE (Common Toxicity Criteria for Adverse Effects) v4.03 will be used.
Overall survival | 2 years
  The number of subjects alive at two years from the first day of salvage therapy.

SECONDARY OUTCOMES:
The number of subjects with a complete response (CR). | Up to Day 60
  A complete response will be defined as bone marrow blasts <5% with absolute neutrophil count ≥1000/μL and platelet ≥100,000/μL.
The number of subjects with CR with incomplete hematologic recovery (CRi) | Up to Day 60
  CRi is defined as CR without platelet recovery or neutrophil recovery. This will be defined as bone marrow blasts <5% with absolute neutrophil count <1000/L and platelet <100,000/L.
The number of subjects in a morphologic leukemia-free state (MLFS). | Up to Day 60
  MLFS is bone marrow blasts <5% with absolute neutrophil count <1000/μL AND platelet <100,000/μL.
The number of subjects experiencing partial remission. | Up to Day 60
  Partial remission (PR) is defined by a decrease of at 50% or more in the percentage of blasts to less than 25% in the bone marrow. and normalized blood counts ( ANC>1000, Platelets>100,000/ml).
Progression-free Survival | 1 Year
  The number of subjects, who from the first day of remission until one year, do not relapse or progress.

CONTACTS AND LOCATIONS:
Overall Officials: Sameem Abedin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwuakee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No